CLINICAL TRIAL: NCT04988828
Title: The Effects of Whole Body Vibration Therapy on Increasing Quadriceps Strength Prior to Anterior Cruciate Ligament Reconstruction
Brief Title: The Effects of Whole-body Vibration on Increasing Quadriceps Strength in Patients With ACL Ruptures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Jihong Qiu, PrincipL Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CREC2019.488
Record Dates: First submitted 2021-07-03; First posted 2021-08-04 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Anterior Cruciate Ligament Injuries; Quadriceps Muscle Atrophy
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): deep squat
  1min*6repetitions
  Interventions: Device: Whole body vibration
- Whole body vibration group (Experimental): deep squat on a whole body vibration platform with 30Hz and 4mm amplitude
  1min*6repetitions
  Interventions: Device: Whole body vibration

INTERVENTIONS:
Device: Whole body vibration — vertical vibration platform with the frequency of 30Hz, amplitude of 4mm. The intervention will last for 5 weeks, twice /week.

SUMMARY:
Introduction: Approximately 35% patients can not return to sports after anterior cruciate ligament reconstruction(ACLR). Persistent quadriceps weakness is a factor that prevents patients return to sports. Pre-operative quadriceps strength is a predictor for the outcomes after ACLR. Therefore, enhancing pre-operative quadriceps is important. However, current prehabilitation can not well restore quadriceps strength may be due to quadricep inhibition. Whole body vibration was proposed as a promising intervention to increase muscle strength and modulate quadriceps inhibition simultaneously. Therefore, this study aim to investigate if whole body vibration has the efficacy of enhancing pre-operative quadriceps and modulating quadricep inhibition in patients with ACL injuries.

Methods: A randomized controlled trial was designed. Patients with primary ACL injuries, age from 18-45 yrs, BMI<29, physically active who awaiting ACLR will be included. Patients with any previous lower-limb injuries within 1 year, any cardiovascular or metabolic disorders will be excluded. All the subjects in this study have to finish their routine 5 week prehabilitation as well as the interventions. The primary outcomes of this study include quadriceps strength and quadriceps central activation ratio. Secondary outcomes include the score of IKDC and ACL-RSI, as well as the concentrations of myokines in serum.

DETAILED DESCRIPTION:
The effect of whole body vibration therapy on increasing quadriceps strength prior to anterior cruciate ligament reconstruction

1. Introduction:

   Anterior cruciate ligament (ACL) injury is a common knee injury in orthopaedic and sports medicine. It is estimated that there are 200000 ACL injuries annually in US. According to the ACL injury registry system of Scandinavia, the incidence of ACL injury was about 32-38/10000 people per year. ACL reconstruction (ACLR) has been recommended as the optimal treatment to restore knee passive laxity in patients with ACL injury who have desire to return to sports. However, a recent meta-analysis showed that only 42% of elite athletes are able to return to non-elite competitive sports following a successful reconstruction and rehabilitation. About 50% of them cannot return to sports at 1 year and one-third cannot return at 2 years post-operatively.

   Until now, the reason why some patients can have good functional recovery following surgery while the others cannot is still unknown. Since the ultimate goal of ACL reconstruction is to help patients return to pre-injury activity without high re-injury risk, identifying those who are at high risk of poor recovery following surgery is extremely essential. Some previous studies concluded that pre-operative quadriceps strength is a key predictor for functional recovery post-operatively. Therefore, increasing pre-operative quadriceps strength is very important. Several studies implemented pre-operative rehabilitation found that part of patients still could not achieve symmetrical quadriceps strength, which mainly because of injury-induced arthrogenic inhibition and increased atrophy-related biomarkers makes those patients have low response to traditional strength training.

   It has been demonstrated that whole body vibration is an effective way in decreasing AMI due to increase corticomotor excitability. Whole body vibration becomes more and more popular as an additional program of physiotherapy for diverse disorders. For patients with ACL injury, previous studies indicate that whole body vibration is effective in improving quadriceps function, neuromuscular control and balance. There are several mechanisms can explain the benefits whole body vibration therapy brought to ACLD patients. Firstly, vibratory stimuli can increase the excitability of type Ia afferent neuron via muscle spindles, resulting in tonic vibration reflex and enlargement of type I and type II muscle fibers. Secondly, whole body vibration can decrease fast-twitch motor unit recruitment thresholds immediately, leading to higher activation of muscles. Thirdly, vibratory stimuli may activate proprioceptive receptors of lower limbs. On molecular level, Low-amplitude high frequency vibration can down regulate Atrogin-1 mRNA and myostatin expression. In addition, it also was found effective in increasing circulating irisin which is a recently identified myokine levels acutely after vibration exercises. Several studies also reported that whole body vibration training can reduce blood concentration of TNF-αreceptors, TNF-α, IL-6 in elderly population and healthy people after exercise. Based on the above, whole body vibration maybe a more efficient and effective way to improve quadriceps strength prior to surgery.

   Thus, this study is primarily to answer the research question: Do patients with greater quadriceps strength improvement prior to surgery also have better functional recovery following ACLR? The second aim is to answer the research question: Are quadriceps inhibition and altered exercise-induced myokines secretion the reasons for the patient's different responses to the same intensity exercise? The third aim is to answer is whole body vibration is a more effective and efficient way to improve quadriceps strength prior to surgery?
2. Methodology:

   A randomized control trial 2.1 Participants: Inclusion criteria: Adult; primary unilateral ACL rupture; no other injuries on lower extremities; BMI <30; no acute symptoms of injury; waiting for ACLR Exclusion criteria: BMI≥ 30; pregnancy; any cardiac or respiratory disease; refuse to accept ACLR 2.2 Interventions: Patients will be randomized allocated into 2 groups: conventional group and; vibration group; conventional+ strength training group; conventional +vibration group.

   Conventional group： strength training Vibration group: Whole body vibration therapy Conventional+ vibration group: strength training+ whole body vibration therapy Strength training protocol: Leg press 75% RM 10 repetitions*3 Leg extension 75% RM 10repetitions*3 Leg curl 75%RM 10 repetitions*3 Hip abduction 75% RM 10 repetitions*3 Hip adduction 75% RM 10 repetitions*3 Straight leg raise 75 RM 10 repetitions*3 Squat 1 min*6 repetitions ,1 min rest between each Whole body vibration (Fitvibe Excel Pro) protocol: Vertical direction vibration Position: standard squat with knee 60 flexion, barefoot and hands on the wrist Frequency: 20-60 Hz (adjusted with a step of 5Hz) Amplitude: 2-4mm Intensity: 15-30 mins (adjusted according to patients' self-reported feeling and progress)

   All of the interventions will take fivefour weeks and patients need to complete 10 sessions of exercise at least.

   In order to make all of the patients follow a same post-operative rehabilitation. A smart phone APP illustrating our post-operative rehabilitation protocol will be installed to patients' smart phones.

   2.3Outcomes: 2.3.1 Time points for outcome measurements: baseline, after a single session of WBV, pre-operation, 3 months post-operation, 9months post-operation.

   2.3.2 Quadriceps strength and quadriceps voluntary activation : Subjects' quadriceps peak torque (both legs) measurement will be completed on an isokinetic strength dynamometer (Biodex System 3, Biodex Medical Systems, Shirley, NY, USA). During the test, subjects are positioned with their hip flexed 90°and knee flexed 30°and subjects are asked to try their very best to ensure the MVIC. Meanwhile, the tester will give encouraging word 'harder and harder' during the process of contraction. The MVIC test will repeat 3 times per subject. And sufficient rest is allowed during the interval of each repeat. In order to standardize the data, individual MVIC peak torque will be divided by the body mass of every subject for the further statistic analysis.

   To quantify quadriceps activation ratio the superimposed burst technique will be used.

   The peak torque recorded from the MVIC test will be inputted into a software to deliver a supramaximal electrical stimulus (from DS7R:10-pulses, 100 Hz train) to the quadriceps muscle once the maximal knee extension torque is reached. The electrical stimulus will be delivered through two self-adhesive stimulating electrodes (8 × 13cm) applied over the vastus lateralis muscle proximally and the vastus medialis distally. Quadriceps activation ratio will be calculated using the central activation ratio formula (CAR), which is (MVIC) / (peak torque generated by the stimulus) *100. A CAR of 100 was used to represent complete quadriceps activation. CAR values that were ≥ 95 were considered to be 'normal' and/or representative of a healthy CAR value. The maximal CAR value that is collected will be used for statistical analysis.

   CAR= MVIC/(MVIC+ST) *100%

   2.3.3 Quadriceps thickness: Previous studies have confirmed that quadriceps size could be accurately predicted from a single MRI scan at the middle level of the thigh. In this study, considering the cost-inefficiency of MRI examination, shear-wave elastography ultrasound (version 6.0; Supersonic Imagine, Aix-en-Provence, France) will be used to estimate quadriceps CSA since several studies demonstrate that ultrasound is a reliable tool for quantification of muscle CSA. Furthermore, Abe T et al. found there is a high correlation(r=0.91) between muscle thickness and CSA of quadriceps. And Franchi et al. support the use of ultrasound-measured middle level quadriceps thickness for monitoring long-term hypertrophic response induced by resistant strength training as an alternative to the much more expensive MRI examination.

   2.3.4 Functional performance (sSingle leg hop; postural control): The single leg hop (SLH) test will be performed as previous studies reported. Before testing, patients will be required to complete a 5 min warm-up on a stationary exercise bike. A general instruction about the jumping task "Stand on one leg, jump as far possible and land on the same leg" will be given. Three trials will be performed with each leg followed by familiarization. The SLH will be deemed correctly if the patient is able to achieve maximal hop distance while maintaining balance for at least 2 s after landing. Patients will be asked to start with their non-injured leg.

   The Biodex Stability System (with software version 3.1, Biodex Medical Systems) will be used to evaluate postural control. Participants will be positioned with both feet on the platform and in a comfortable position with knee flexion around 15°. The foot positions recorded in the first session will be used at all subsequent assessments. Each patient have to maintain the static position with the platform progressively decreased in stability from level 8 to level 4 within 25 seconds. There will be a total of 3 trials, with a 10-second resting time between. The mean ±standard deviation of the OSI, API, and MLI will be recorded.

   2.3.5 Patients reported outcomes: The subjective functional outcome will be evaluated by Lysholm knee scoring system, the IKDC subjective scoring system and Tegner activity score. Psychological readiness for return-to-play will be evaluated by ACL-RSI. The IKDC is consisted of 10 questions about symptoms and activity ranging from 0 to 100 where 100 implies perfect knee function. The Tegner score is an activity level scaled from 1 (low activity) to 10 (very high activity). The ACL-RSI scale with 12 items measures three specific psychological constructs-emotions, confidence in performance and risk appraisal-on a scale from 0 to 100. This scale is a predictive parameter for a successful RTS after ACLR.

   2.3.6 Biomarkers in blood serum: Blood will be taken at baseline, at 30 mins after 1 day exercises and when after completion 4 weeks exercises.

   The technique for serum sampling was reported by Perez-Lopez et al . Blood samples will be centrifuged for 15 minutes at 1000 g and stored at -80°C. Two high-sensitivity enzyme-linked immunosorbent assay (ELISA) kits will be used to determine the serum concentration of IL-15, IL-15Rα, myostatin, IL-6, IL-10, IGF-1, irisin in duplicates.

   2.3.7 Swelling and pain assessment: (will be measured 1 week and 3 months post-operatively) Knee joint swelling will be evaluated by measurement of mid-patellar girth with a standard tape measure (tape width = 8 mm). Difference between injured side and contralateral side will be recorded for further analysis. The same experienced researcher will perform the measurement.

   Pain will be estimated by the well-established numerical pain rating scaleThe well-established numerical pain rating scale will estimate pain. Patients will finish this scale based on their subjective feeling according to the introduction on the scale.

   2.3.8 Knee passive laxity The knee passive laxity will be measured by KT-1000 knee arthrometer. The KT-1000 is an objective instrument for ACL injury and reconstruction, which measures anterior tibial motion relative to the femur. The test involves strapping the KT-1000 to the leg, pulling the tibia anteriorly, and quantifying the amount of movement in millimeters (mm).

   2.3.9 Motivation and Social Cognitive Variable and Rehabilitation Adherence For measuring treatment motivation, the injury rehabilitation version of Treatment Self-Regulation Questionnaire will be used. The questionnaire has been used among ACL patients in Hong Kong and has received supporting evidence for its validity and reliability. For measuring the variables from the theory of planned behaviour, the Chinese injury rehabilitation version of the Theory of Planned Behaviour Scale that has been developed and validated from previous studies about injury rehabilitation will be used .

   The rehabilitation adherence will be estimated by the Self-Reported Injury Rehabilitation Adherence Scale. The scale is one of the most widely used self-reported instrument that has been validated in Chinese language, and it has also been used among ACL patients for measuring their rehabilitation adherence with strong evidence to support its psychometric properties.
3. Statistics:

Quadriceps strength was used as the primary outcome. With an estimated effect size of 0.3 for the increase in quadriceps strength after WBV based on a similar study and assuming a 20% attrition rate, it was demonstrated that each group should recruit 50 subjects, and 125160 in total. Baseline characteristics will be tested using independent t tests for parametric parameters and the x2 test for nonparametric parameters. Repeated-measures analysis of variance (ANOVA) with time as the repeated-measures factor for the outcomes measure will be used to analyze the difference between the 24 groups. Tests of within-patient effect were utilized to find any difference between different time intervals in each group. Contrast with F statistics will be used to detect the difference at different time points in the post hoc analysis. The Mann-Whitney U test will be employed to compare for any difference between the 24 groups in the outcome variables. For all statistical tests, the alpha level will be set at 0.05 and performed using the Statistical Package for Social Sciences (IBM SPSS Ver. 24).

ELIGIBILITY:
Inclusion Criteria:

* BMI<19
* ACL injuries
* no previous lower limb injury within 1 year
* physically active before the injury

Exclusion Criteria:

* pregnant
* have any cardiovascular
* nervous or metabolic disorders

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
quadriceps strength | change from baseline to finishing the intervention
  Subjects' quadriceps peak torque (both legs) measurement will be completed on an isokinetic strength dynamometer (Biodex System 3, Biodex Medical Systems, Shirley, NY, USA). During the test, subjects are positioned with their hip flexed 90°and knee flexed 30°and subjects are asked to try their very best to ensure the MVIC. Meanwhile, the tester will give encouraging word 'harder and harder' during the process of contraction. The MVIC test will repeat 3 times per subject. And sufficient rest is allowed during the interval of each repeat. In order to standardize the data, individual MVIC peak torque will be divided by the body mass of every subject for the further statistic analysis.
quadriceps central activation ratio | change from baseline to finishing the intervention
  he peak torque recorded from the MVIC test will be inputted into a software to deliver a supramaximal electrical stimulus (from DS7R:10-pulses, 100 Hz train) to the quadriceps muscle once the maximal knee extension torque is reached. The electrical stimulus will be delivered through two self-adhesive stimulating electrodes (8 × 13cm) applied over the vastus lateralis muscle proximally and the vastus medialis distally. Quadriceps activation ratio will be calculated using the central activation ratio formula (CAR), which is (MVIC) / (peak torque generated by the stimulus) *100. A CAR of 100 was used to represent complete quadriceps activation. CAR values that were ≥ 95 were considered to be 'normal' and/or representative of a healthy CAR value. The maximal CAR value that is collected will be used for statistical analysis.

SECONDARY OUTCOMES:
International Knee Documentation Committee Subjective Knee Form (IKDC) | change from baseline to finishing the intervention
  The IKDC is consisted of 10 questions about symptoms and activity ranging from 0 to 100 where 100 implies perfect knee function.
Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) | change from baseline to finishing the intervention
  The ACL-RSI scale with 12 items measures three specific psychological constructs-emotions, confidence in performance and risk appraisal-on a scale from 0 to 100. In this scale, higher score indicates better psychological readiness of patients to return to sports.
International Physical Activity Questionnaire - Short Form (IPAQ) | Every week during the 5 week interventions
  This measure assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting. The specific types of activity that are assessed are walking, moderate-intensity activities and vigorous intensity activities; frequency (measured in days per week) and duration (time per day) are collected separately for each specific type of activity. These following values continue to be used for the analysis of IPAQ data: Walking = 3.3 METs, Moderate PA = 4.0. There is no exact range of the IPAQ score. In addition, higher scores mean more active lifestyle and higher intensity of daily activity.
  METs and Vigorous PA = 8.0 METs.

CONTACTS AND LOCATIONS:
Overall Officials: Michae Tim-Yun Ong, MSc, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince Wales Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Qiu J, Ong MT, Choi CY, Cao M, Ko VM, He X, Fu SC, Fong DTP, Yung PS. Five Weeks of Whole-body Vibration in Prehabilitation for Knee Function Following Anterior Cruciate Ligament Reconstruction: A Single-blinded Randomized Controlled Trial. Sports Med Open. 2025 Aug 22;11(1):98. doi: 10.1186/s40798-025-00901-1. PMID 40844690